CLINICAL TRIAL: NCT06505993
Title: COVID19 -- Health Communication and Structural Intervention Evaluation -- K-VAC: Kentucky Vaccinating All Communities
Brief Title: Addressing COVID-19 Vaccine Hesitancy With Muliti-Level Interventions in Appalachia
Acronym: K-VAC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Kiviniemi (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Marc Kiviniemi, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 88486; R01MD016864 (NIH)
Record Dates: First submitted 2024-07-16; First posted 2024-07-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Vaccine Hesitancy
Keywords: COVID-19; Multi-Level Intervention; Vaccine Hesitancy; Rural
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Health Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Health Communication (Experimental): This intervention arm will include exclusively health communication messaging strategies that is both theory-based and community-targeted to encourage uptake of the COVID-19 vaccine delivered by trusted local communicators. Pre-identified theory-based components are attitudes, social norms, perceived behavioral control, response efficacy, and implementation intentions. The development process for the messaging will be based through a conjoint process of identification of theory- based determinants of decision-making relevant to the desired behavior change and a community-engaged process of identifying: a) community-specific messaging themes; b) trusted communicators within the target population; and c) community-specific messaging, imaging, and themes to achieve targeting.
  Interventions: Behavioral: Health Communication
- Health Communication + Structural (Experimental): This intervention arm will include the conditions outlined and included in the health communication arm, however, they will be coupled with a series of structural and/or environmental intervention strategies as well, which are targeted to facilitate vaccine accessibility and uptake among adults in the randomly assigned study counties.
  Interventions: Behavioral: Health Communication + Structural
- Standard of Care (No Intervention): No study-specific intervention strategies (as outlined above) will be implemented in control counties at the time of the study period. Any ongoing and/or pre-existing efforts within the scope of the project's outcomes will continue as it would have i.e. a health department operating a health fair.

INTERVENTIONS:
Behavioral: Health Communication — Participants will experience a coordinated social marketing campaign including targeted messaging related to vaccine education, self-efficacy, and informative resources to receive the COVID-19 vaccine. The intervention messaging will be strategically layered and disseminated to this intervention arm predominately via Facebook by trusted and local communicators in the study counties.
  Arms: Health Communication
Behavioral: Health Communication + Structural — This multi-level intervention will include the defined health messaging intervention components, as well as a combination of structural-level intervention strategies targeted to better facilitate access to community-based vaccination delivery. Health organizations will receive a toolkit, which will include community-specific resources and training modules such as: up to date evidence-based vaccination guidance that can be delivered to patients; strategies for navigating conversations with patients about vaccination; any applicable reimbursement, insurance, or qualifying enrollment information specific to the healthcare organization; identifying locations that facilitate access for the community members; provided advertising to promote the locations and timing of the vaccinations; and generating community-based branding for all vaccination delivery based on the trusted information sources identified.
  Arms: Health Communication + Structural

SUMMARY:
The purpose of this community-engaged study is to test the ability of county-level strategies to increase uptake of COVID-19 vaccination. In this study the key objective is to test whether health communication strategies or health communication + county-specific structural/environmental support increases COVID-19 vaccine uptake and changes perceptions and beliefs about the vaccination at the county-level.

DETAILED DESCRIPTION:
The intervention trial will be a community-based, three-arm cluster randomized controlled trial. The three arms are: (1) multilevel invention (vaccine communication campaign + community-level structural intervention),(2) health communications only intervention, and (3) control/standard of care. Randomization will take place at the county level. The 15 participating counties will first be matched into blocks of three, with each block being matched as closely as possible on recent county influenza vaccination rates. After matching, the three counties within each matched block will be randomly assigned to one of the three study arms. This technique of randomizing to study arm within each matched block of counties increases confidence that community-level factors that might influence vaccine uptake are equally distributed across study arms. Following randomization, the intervention process will begin in counties in the multilevel and communication campaign intervention arms. Assessment of primary and secondary study outcomes will take place 6 months after initiation of the intervention. Finally, after assessment of outcomes is complete, the intervention components will be offered to the control counties.

ELIGIBILITY:
Up to 2,250 participants will take part in the study --- approximately 150 residents in each of the 15 participating Appalachian Kentucky Counties. In each of the fifteen counties, the investigators will collect survey data from 150 adults who are served by Homeplace, a medical and social services organization run by the UK Center for Excellence in Rural Health, which provides services in each of the 15 partner counties. Homeplace provides services to adults who are medically underserved and typically at 100-133% of the federal poverty level, primarily through service delivery by trained local Community Health Workers (CHWs). CHWs will recruit participants and collect the survey data from the identified individuals. Importantly, the criteria for qualification for Homeplace services are equivalent across the 15 counties, providing equivalence of sample across counties. A random sample of 150 individuals per county will be drawn from the Homeplace client database for that county. Gender, ethnic background, and health status will roughly mirror that of the demographics of the county.

Inclusion Criteria:

1. Must be a current Homeplace client
2. Live in one of the 15 selected study counties
3. Over the age of 18
4. Have the ability to complete the survey in English

Exclusion Criteria:

1. Not a current Homeplace client
2. Primary residence is not in one of the 15 study counties
3. Not within the ages of 18-99 years old
4. English is not your primary language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccination uptake | Baseline and 6 months
  Change in *county-level* vaccination rates- to assess uptake, the investigators will ascertain the number of individuals in each county who received the COVID-19 vaccination during the intervention period as well as during an equivalent time frame prior to the intervention. This assessment will be obtained from existing, deidentified vaccination rate data maintained by the KY Department of Public Health. The primary outcome variable will be the number of individuals receiving vaccination.

SECONDARY OUTCOMES:
COVID-19 Vaccination Behaviors | Baseline and 6 months
  The investigators will assess individual-level vaccination behaviors with a survey among adults in each study county. To capture, participants will be asked to self-report their responses to following statements with multiple choice answer choices provided to allow for quantitative analysis: 1) "Have you or do you think you have had COVID-19?" 1= Yes I was tested or a doctor diagnosed me; 2= Maybe I had some symptoms but was not tested; 3= No. 2) "How many times have you had COVID-19?" 1= Once, 2= Twice, 3= Three or more times. Additionally, the investigators will use a 4-point Likert scale (1= strongly disagree, 2= disagree, 3= agree, 4= strongly agree) to assess respondent likeliness of intention to vaccinate with either a COVID-19 booster, or COVID-19 vaccine, in the next 12-months.
COVID-19 Attitudes | Baseline and 6 months
  The investigators will assess individual-level vaccination attitudes and beliefs with a survey among adults in each study county. Participants will be asked to self-report their responses to following statements utilizing a 4-point Likert scale (1= strongly disagree, 2= disagree, 3= agree, 4= strongly agree):
  1. "I feel safe about getting the COVID-19 vaccine."
  2. "The COVID-19 vaccine may cause short term problems, like fever or discomfort."
  3. "The COVID-19 vaccine is being pushed to make money for drug companies."
  4. "The COVID-19 vaccine was not tested enough for safety."
  5. "The COVID-19 vaccine may cause lasting health problems."
  6. "I am concerned that the COVID-19 vaccine will cost more than I can pay."
  7. "The COVID-19 vaccine was developed too quickly."
COVID-19 Risk Perceptions | Baseline and 6 months
  The investigators will assess individual-level risk perceptions about vaccination with a survey among adults in each study county. Participants will be asked to self-report their responses to following questions with a 4-point Likert scale:
  1. "How likely are you to get COVID-19 in the next 6 months?" 1= very unlikely to 4= very likely
  2. "How afraid are you of getting COVID-19 in the next 6 months?" 1= not afraid at all to 4= extremely afraid
  3. "If you were to get COVID-19 in the next 6 months, how serious would it be?" 1= not serious at all to 4= extremely serious

CONTACTS AND LOCATIONS:
Overall Officials: Marc T. Kiviniemi, PhD, Principal Investigator — University of Kentucky; Kathryn M. Cardarelli, PhD, MPH, Principal Investigator — University of Louisville
Locations (1):
- University of Kentucky Center of Excellence in Rural Health, Hazard, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No